CLINICAL TRIAL: NCT06081504
Title: Wii Fit Exercises Versus Pilates Exercises on Muscle Strength, Postural Balance, and Functional Performance in Adult Patients With Lower Extremity Burn
Brief Title: Wii Fit Exercises Versus Pilates Exercises in Adult Patients With Lower Extremity Burn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ahmed Elsayeh, Lecturer of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004387
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Burns; Muscle Weakness; Exercises; Functional Performance
Keywords: Wii Fit exercises; Pilates exercises; muscle strength; postural balance; functional performance; lower extremity burn
MeSH Terms: conditions — Burns; Muscle Weakness; Motor Activity

STUDY DESIGN:
Intervention Model Description: Forty-five patients of both sexes with healed LL burns will be allocated randomly into three groups: the Wii fit exercises group, the pilates exercises group, and the standard physical therapy group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wii fit exercises group (Experimental): Fifteen patients will be engaged in the Wii Fit exercises program for 30 minutes in addition to the standard physical therapy program, 3 sessions a week for 12 weeks.
  Interventions: Other: Wii fit exercises program; Other: Standard physical therapy program
- Pilates exercises group (Experimental): Fifteen patients will be engaged in the Pilates exercises program for 30 minutes in addition to the standard physical therapy program, 3 sessions a week for 12 weeks.
  Interventions: Other: Pilates exercises program; Other: Standard physical therapy program
- Standard physical therapy group (Active Comparator): Fifteen patients will be engaged in the Standard physical therapy program (lower limb stretching and strengthening exercises and deep friction massage) for 45 minutes, 3 sessions a week for 12 weeks.
  Interventions: Other: Standard physical therapy program

INTERVENTIONS:
Other: Wii fit exercises program — Wii fit exercises for balance training and lower limb strengthening for 30 minutes. In addition to warming up and cooling down, 10 minutes each in the form of a range of motion exercises and stretching.
  Arms: Wii fit exercises group
Other: Pilates exercises program — Selected pilates exercises for balance training and lower limb strengthening: Articulating bridge, Spine stretch, Single leg stretch, Double leg stretch, Criss-cross, One leg kick, Side kick, Hip twist, and Standing footwork for 30 minutes, 10 repetitions each. In addition to the warming up and the cooling down exercises before and after the pilates exercises, 10 minutes each in the form of a range of motion exercises and stretching, and deep friction massage for scar management.
  Arms: Pilates exercises group
Other: Standard physical therapy program — All patients will receive the standard physical therapy program consisting of 45 minutes per session of a supervised and individualized exercise program for three sessions per week for eight weeks which will include: Stretching exercises for lower limb muscles, each stretch will be maintained for 45 seconds, 3 repetitions, strengthening exercises for lower limb muscles starting from 50 to 60% of 1 repetition maximum and the intensity will be increased gradually until 80 to 85 % through the treatments weeks.

SUMMARY:
The aim of the study is to compare the effect of Wii fit exercises and Pilates exercises on muscle strength and postural balance, and functional performance in adult patients with lower extremity burn.

DETAILED DESCRIPTION:
Severe burn injuries are associated with hypermetabolic response and increased catabolism. These lead to a vast loss of muscle mass and reduced muscle strength. The main concern of burn injury rehabilitation has shifted from survival to optimizing functional outcomes and speeding up work return. Lower limbs (LL) are considered the most burned body parts, resulting in many potential complications, including pain, contractures, scars, altered sensations, muscle weakness, and postural balance impairment.

Video game systems are more cost-effective than developing custom-designed rehabilitation equipment and are becoming increasingly popular among individuals undergoing physical rehabilitation. Among the most common video game systems used for this purpose (Wii Fit, Dance Revolution, EyeToy, and Kinect), Nintendo's Wii Fit is the most popular. It was the first video game system to use body movements as a game controller. The exerciser stands on an external balance board and controls the movement of a virtual character in the game by changing the center of pressure on the board. The game provides both visual and auditory feedback to the exerciser. This system combines fun with physical exercise for all ages as it allows for work on joint flexibility, muscular strength, and postural ergonomics.

Pilates is a mind/body exercise that requires core stability, strength, flexibility, and attention to muscle control, posture, and breathing. Pilates exercise is performed solo in one's own space, so there is no risk of collision or other contact with others. The risk of injury to the musculoskeletal system is therefore minimized, making Pilates a relatively safe form of exercise.

To the authors' knowledge there are no previous studies comparing the effect of Wii fit exercises and Pilates exercises on muscle strength and postural balance, functional performance in adult patients with lower extremity burn so, this study is designed to compare the effect of Wii fit exercises and Pilates exercises on muscle strength and postural balance, functional performance in adult patients with lower extremity burn.

ELIGIBILITY:
Inclusion Criteria:

* The patients' age will range from 35 to 55 years.
* The patients' weight range is from 60 to 85 kg and their height ranges from 155 to 170 cm.
* The total burned surface area (TBSA) is more than 40% measured by the rule of nine.
* Patients with thermal burn only, partial-thickness burn injury, and at least 3 months after burn injuries.
* Patients with low physical activity levels.

Exclusion Criteria:

* Patients with inhalation injury.
* Patients with leg amputation.
* Patients with any limitation in lower limb range of motion.
* Patients with auditory or visual problems.
* Patients with congenital musculoskeletal deformities, especially in the foot.
* Patients with psychiatric disorders.
* Patients with lower limb paralysis.
* Patients with cardiac abnormalities or cardiac pacemakers.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-11 (Estimated)

PRIMARY OUTCOMES:
Isokinetic Muscle Strength Assessment | Change from baseline at twelve weeks after the intervention
  Isokinetic Muscle Strength Assessment will be assessed by A Biodex dynamometer (Biodex Medical System, Shirley, NY, USA). The values of knee flexors and extensors muscle peak torque of dominant leg were measured regardless the location of burns at an angular velocity of 150°/seconds, hip angle of 100° and patient were supported with a securing belt placed over the mid- thigh, pelvis and trunk. Three sub-maximal repetitions were allowed for the patient without any load as a warm-up. The patient then carried out 10 of maximum voluntary muscle contractions continuously without rest and the highest values were recorded for analysis.
Dynamic balance score | Change from baseline at twelve weeks after the intervention
  The dynamic balance score will be measured by the Biodex Balance System (Biodex Medical System, Shirley, NY, USA). The Biodex Balance System is a valid and reliable method to assess dynamic balance.
  A Biodex Balance System (Biodex Medical Systems, Shirley, NY) consists of a movable balance platform that provides a 20° surface tilt through a 360° range of motion. The platform interfaces with computer software that enables the device to serve as an objective assessment of balance. All measurements were performed at level eight of stability, and the test duration was set at 20 seconds for three successive trials

SECONDARY OUTCOMES:
Functional exercise capacity | Change from baseline at twelve weeks after the intervention
  Six-minute walk test will be used to assess functional exercise capacity of the participants. The 6-MWT was performed in a 30-meters flat corridor according to the American Thoracic Society guidelines. Patients were asked to walk as far as possible in the 30-m corridor during the 6-min period. Standardized verbal encouragement is given to the patients during the 6-MWT. At the end of the test, the walking distance was measured. The predicted values of 6-MWT were calculated according to age and gender

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa MA El Sayeh, Principal Investigator — Lecturer at Faculty of Physical Therapy, Cairo University
Locations (2):
- Egypt (2):
  - Shaimaa Mohamed Ahmed El Sayeh, Cairo, New Cairo
  - Shaimaa Mohamed Ahmed El Sayeh, Cairo

IPD SHARING:
Plan to Share IPD: No